CLINICAL TRIAL: NCT00611130
Title: Vigabatrin for Treatment of Cocaine Dependence: A Phase II Study
Brief Title: Vigabatrin for Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPP-01004
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Addiction; Dependence; Treatment
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 3 Vigabatrin Tablets, 500 mg, bid, for 9 weeks
  Interventions: Drug: vigabatrin
- 2 (Placebo Comparator): 3 Placebo Tablets, bid, for 9 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vigabatrin — Tablets twice a day for 9 weeks
  Other Names: CPP-109, VGB, GVG
  Arms: 1
Drug: placebo — tablets twice daily for 9 weeks
  Arms: 2

SUMMARY:
The objective of this study is to demonstrate that a larger proportion of vigabatrin-treated subjects than placebo-treated subjects will be cocaine-free in the last 2 weeks of treatment.

DETAILED DESCRIPTION:
Cocaine addiction, a serious public health concern associated with significant medical, social, and economic consequences, is difficult to treat using traditional psychosocial and behavioral therapies. Despite testing of a number of different agents for cocaine dependency, there remains no proven pharmacologic treatment for cocaine addiction.

The addictive properties of cocaine have been associated with its actions on mesotelencephalic dopamine reward pathways in the central nervous system (CNS). Cocaine administration increases the levels of dopamine, a neurotransmitter associated with sensations of pleasure and reward. Therefore, blocking cocaine-induced increases in dopamine levels represents a valid pharmaceutical approach to the treatment of cocaine addiction.

Another neurotransmitter, gamma-aminobutyric acid (GABA), suppresses striatal dopamine release, and attenuates cocaine-induced increases in extracellular and synaptic dopamine levels in the striatum and nucleus accumbens in animal models of drug dependence. Significant elevation of brain GABA levels may reduce cocaine-stimulated dopamine release and dampen the sensations of pleasure and reward. Thus, drugs that potentiate or enhance GABA-ergic transmission are candidates for the treatment of cocaine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and provide written informed consent.
* Male or female at least 18 years of age.
* Meets DSM-IV (Diagnostic and Statistical Manual of Mental Disorders Fourth Edition) criteria for cocaine dependence as primary diagnosis, as determined by the Substance Abuse module of SCID (Structured Clinical Interview for DSM-IV).
* Provide at least one urine sample that is positive for cocaine according to a rapid screening test.
* Seeking treatment for cocaine dependence.
* Have normal visual fields.
* Be in generally good health based on history, physical examination, electrocardiogram and laboratory findings.
* If female of childbearing potential, use acceptable contraceptive methods. (oral contraceptives (the pill), IUDs, contraceptive implants under the skin, contraceptive rings or patches or injections, diaphragms with spermicide, and condoms with spermicide). Surgical sterilization by tubal ligation or hysterectomy is acceptable

Exclusion Criteria:

* Has current dependence, as determined by the SCID, on any psychoactive substance other than cocaine, alcohol, nicotine, or marijuana or physiologic dependence on alcohol requiring medical detoxification.
* Has any serious medical or psychiatric illness and/or clinically significant abnormal laboratory value, which in the judgment of the Principal Investigator or his/her designee would make study participation unsafe, or would make treatment compliance difficult or put the study staff at undue risk.
* Be under court mandate to obtain treatment.
* Be enrolled in an opiate substitution treatment program within 2 months of randomization.
* Has ever taken vigabatrin in the past.
* Is pregnant or lactating.
* Has clinically significant ophthalmologic disease, which would preclude safety monitoring or is undergoing treatment for ocular disease.
* Has received a drug with known major organ toxicity, including retinotoxicity within 30 days of randomization.
* Is currently participating in, or has been enrolled in another clinical trial within the last 30 days.
* Be anyone who, in the judgment of the investigator, would not be expected to attend regular study visits or to complete the study protocol, due to imminent relocation from the clinic area, legal difficulties, work-related problems, transportation, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, MD, PhD, Principal Investigator — University of Cincinnati
Locations (11):
- United States (11):
  - Addiction Treatment Clinic, Little Rock, Arkansas
  - St. Luke's Hospital Addiction Pharmacology Research Laboratory, San Francisco, California
  - Friends Research Institute, Torrance, California
  - Operation PAR, Largo, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Johns Hopkins Bayview Medical Center Center for Chemical Dependence, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - New York University Mental Health and Addictive Disorders Research Program, New York, New York
  - Cincinnati Addiction Research Center (CinARC), Cincinnati, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Somoza EC, Winship D, Gorodetzky CW, Lewis D, Ciraulo DA, Galloway GP, Segal SD, Sheehan M, Roache JD, Bickel WK, Jasinski D, Watson DW, Miller SR, Somoza P, Winhusen T. A multisite, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of vigabatrin for treating cocaine dependence. JAMA Psychiatry. 2013 Jun;70(6):630-7. doi: 10.1001/jamapsychiatry.2013.872. PMID 23575810
- [Derived] Berezina TL, Khouri AS, Winship MD, Fechtner RD. Visual field and ocular safety during short-term vigabatrin treatment in cocaine abusers. Am J Ophthalmol. 2012 Aug;154(2):326-332.e2. doi: 10.1016/j.ajo.2012.02.026. Epub 2012 Jun 15. PMID 22704138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 01/08-01/09 at 11 US research trial sites.
Pre-assignment Details: After Informed Consent obtained, subjects entered a 2-4 week Screening/Baseline Phase to determine whether all Inclusion/Exclusion Criteria were met. Randomization strata included gender, primary method of cocaine administration (snort or intravenous/smoke) & use in last 30 days (≤18 days or >18 days)
Groups:
- CPP-109 Vigabatrin: CPP-109 tablets, 500 mg. 3 Tablets bid.
- Placebo: Matching Placebo Tablets. 3 tablets bid.
Period: Overall Study
Arm/Group | CPP-109 Vigabatrin | Placebo
Started | 92 | 94
Completed 12 Week Treatment Phase | 61 | 64
Completed | 43 | 47
Not Completed | 49 | 47
Not completed — Lost to Follow-up | 25 | 29
Not completed — Protocol noncompliance | 7 | 6
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Other | 5 | 4
Not completed — Incarceration | 3 | 2
Not completed — Administrative | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPP-109 Vigabatrin | Placebo | Total
Number analyzed (Participants) | 92 | 94 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (7.62) | 45.0 (8.33) | 44.8 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 60 | 64 | 124
Region of Enrollment [Number; unit: participants]
  United States | 92 | 94 | 186

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Group Abstinent During the Last 2 Weeks of Treatment.
Description: Number of subjects in the CPP-109 Vigabatrin Group vs. Number in Placebo Group abstinent from using cocaine during Weeks 11 and 12 of the Treatment Phase.
Time Frame: Week 13
Population: intent-to-treat
Measure: Number; unit: participants
Groups:
- CPP-109 Vigabatrin Tablets, 500 mg: Vigabatrin Tablets, 1.5 g bid po, 12 weeks, computerized cognitive behavioral therapy plus contingency management.Subjects proceeded to a 12 week Treatment Phase, including a 2 week dose escalation period, a 9 week maintenance period (3.0 gm/day of vigabatrin) and a 1 week medication taper period. Finally, subjects then proceeded to a 12 week follow-up period. Subjects attended clinic visits 3 times per week (typically on Monday, Wednesday, and Friday) for efficacy and safety assessments and for treatment during the Screening/Baseline Phase and the 12 week Treatment Phase. Subjects returned for follow up visits at Weeks 13, 16, 20 and 24.
- Matching Placebo Tablets: Subjects proceeded to a 12 week Treatment Phase,receiving 3 tablets bid po Finally, subjects then proceeded to a 12 week follow-up period. Subjects attended clinic visits 3 times per week (typically on Monday, Wednesday, and Friday) during the Screening/Baseline Phase and the 12 week Treatment Phase. Subjects returned for follow up visits at Weeks 13, 16, 20 and 24.
Arm/Group | CPP-109 Vigabatrin Tablets, 500 mg | Matching Placebo Tablets
Number analyzed (Participants) | 92 | 94
participants | 7 | 5

2. Post Hoc Outcome: Medication Compliance
Description: Using retained urine samples and prior to unblinding, up to 12 specimens/ subject were analyzed for vigabatrin levels. Compliance assessment based on > or = 70% of urines in subjects assigned to vigabatrin having quantitative levels of vigabatrin indicaticative of taking drug within the last 24 hours of clinic visit.
Time Frame: Week 2, 4, 6 & 9-11
Population: Completers were defined as those who attended the scheduled Week 13 visit or the third visit of Week 12 and who also had provided urines during Weeks 11 & 12.
Measure: Number; unit: participants
Groups:
- Treatment Phase Completers: Up to 12 urine specimens out of 37 collected during the Treatment Phase completers were analyzed for vigabatrin levels.
Arm/Group | Treatment Phase Completers
Number analyzed (Participants) | 125
participants
  Number of Vigabatrin Completers Analyzed | 61
  Number Medication Compliant | 24

ADVERSE EVENTS:
Groups:
- CPP-109 Vigabatrin Tablets, 500 mg: Vigabatrin Tablets, 1.5 g bid po, 12 weeks. Subjects proceeded to a 12 week Treatment Phase, including a 2 week dose escalation period, a 9 week maintenance period (3.0 gm/day of vigabatrin), and a 1 week medication taper period. Finally, subjects then proceeded to a 12 week follow-up period. Subjects were scheduled for clinic visits 3 times per week (typically on Monday, Wednesday, and Friday) during the Screening/Baseline Phase and the 12 week Treatment Phase. Subjects returned for follow up visits at Weeks 13, 16, 20 and 24.
- Matching Placebo Tablet: Subjects proceeded to a 12 week Treatment Phase,receiving 3 tablets bid po Finally, subjects then proceeded to a 12 week follow-up period. Subjects were scheduled for clinic visits 3 times per week (typically on Monday, Wednesday, and Friday) during the Screening/Baseline Phase and the 12 week Treatment Phase. Subjects returned for follow up visits at Weeks 13, 16, 20 and 24.
Arm/Group | CPP-109 Vigabatrin Tablets, 500 mg | Matching Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 6/92 | 0/94
Other Adverse Events (participants affected / at risk) | 73/92 | 81/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPP-109 Vigabatrin Tablets, 500 mg (N=92) | Matching Placebo Tablet (N=94)
Drug Abuse & Major Depression (Psychiatric disorders) | 2 | 0
Gun shot wound, road traffic accident & tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Hepatitis, acute (Hepatobiliary disorders) | 1 | 0
Meningitis & Pneumonia (Infections and infestations) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPP-109 Vigabatrin Tablets, 500 mg (N=92) | Matching Placebo Tablet (N=94)
Photopsia (Eye disorders) | 8 | 1
Blurred vision (Eye disorders) | 6 | 6
Visual disturbance (Eye disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 14 | 15
Nausea (Gastrointestinal disorders) | 9 | 17
Stomach discomfort (Gastrointestinal disorders) | 3 | 7
Toothache (Gastrointestinal disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 1 | 7
Fatigue (General disorders) | 7 | 9
Nasopharyngitis (Infections and infestations) | 17 | 17
ALT decreased (Investigations) | 7 | 0
CPK increased (Investigations) | 6 | 3
Weight increased (Investigations) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6
Headache (Nervous system disorders) | 10 | 26
Somnolence (Nervous system disorders) | 5 | 5
Dizziness (Nervous system disorders) | 3 | 6
Anxiety (Psychiatric disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 7 | 3

LIMITATIONS AND CAVEATS:
Lack of subject medication compliance, site-to-site variability in medication compliance possibly indicative of differing site capabilities to attract subjects sufficiently motivated to stop using cocaine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days